CLINICAL TRIAL: NCT01759680
Title: Effects of 3 Months of Controlled Whole Body Vibrations With Low Exposure Period on the Risk of Falls Among Nursing Home Residents
Brief Title: Effects of 3 Months of Controlled Whole Body Vibrations on the Risk of Falls Among Nursing Home Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Charlotte Beaudart, PhD Student, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPEES/CB/WBV01
Record Dates: First submitted 2012-12-21; First posted 2013-01-03 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Falls
Keywords: Risk of falls; Whole Body Vibration; Nursing Home

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whole Body Vibration Group (Experimental): The whole body vibration group received 3 training sessions every week composed of 5 series of 15 seconds of vibrations at 30 Hz intensity.
  Interventions: Device: Vibrosphère device
- Control Group (No Intervention): The control group had a normal daily life for the whole study period

INTERVENTIONS:
Device: Vibrosphère device — Vertical Sinusoidal vibration
  Other Names: Whole Body Vibration
  Arms: Whole Body Vibration Group

SUMMARY:
Tiredness, lack of motivation and low compliance can be observed in nursing home residents during the practice of physical activity. Because exercises should not be too vigorous, whole body vibration could potentially be an effective alternative.

The objective of this randomized controlled trial is to assess the impact of 3-month training by whole body vibration on the risk of falls among nursing home residents.

Patients were randomized into two groups: the whole body vibration group which received 3 training sessions every week composed of 5 series of only 15 seconds of vibrations at 30 Hz intensity and a control group with normal daily life for the whole study period.

The impact of this training on the risk of falls was assessed blindly by three tests: the Tinetti Test, the Timed Up and Go test and a quantitative evaluation of a 10-second walk performed with a tri-axial accelerometer.

ELIGIBILITY:
Inclusion Criteria:

* Resident of nursing home
* Able to move

Exclusion Criteria:

* weighing more than 150 kg
* having electronic implants (e.g. pacemaker, brain stimulators)
* having prosthetic hips or knees
* suffering from epilepsy, bleeding disorders, inflammatory abdominal disorders or at high risk of thromboembolism.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Risk of fall | 3 months
  Tinetti test < 19 points = high risk of falls

SECONDARY OUTCOMES:
Risk of fall evaluated by the Timed up and Go test | 3 months
  A timed Up and Go > 14 seconds = high risk of falls
Risk of falls evaluated by the Locometrix | 3 months
  Locometrix is a walking test

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Bruyère, PhD, Study Director — University Of Liège, Department of Public Health, Epidemiology and Health Economics, Liège, Belgiulm
Locations (1):
- University of Liège, Liège, Liège, Belgium

REFERENCES:
- [Derived] Beaudart C, Maquet D, Mannarino M, Buckinx F, Demonceau M, Crielaard JM, Reginster JY, Bruyere O. Effects of 3 months of short sessions of controlled whole body vibrations on the risk of falls among nursing home residents. BMC Geriatr. 2013 May 6;13:42. doi: 10.1186/1471-2318-13-42. PMID 23647914